CLINICAL TRIAL: NCT04379531
Title: Low-dose Computed Tomography in COVID-19 Pneumonia: a Prospective Moscow Study
Brief Title: LDCT in COVID-19 Pneumonia: a Prospective Moscow Study
Acronym: LDCTiP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department (Other)
Responsible Party: Principal Investigator, Sergey Morozov, Chief Research Officer, Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-1
Record Dates: First submitted 2020-04-30; First posted 2020-05-07 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-05

CONDITIONS: Pneumonia; Coronavirus Infection
Keywords: Low-dose CT; Community-acquired pneumonia; Computed tomography
MeSH Terms: conditions — Pneumonia; Coronavirus Infections; Community-Acquired Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Chest CT (Active Comparator)
  Interventions: Diagnostic Test: Low-dose Chest CT
- Low-dose Chest CT (Experimental)
  Interventions: Diagnostic Test: Low-dose Chest CT

INTERVENTIONS:
Diagnostic Test: Low-dose Chest CT — Patients referred by the primary care physician with suspected pneumonia.

SUMMARY:
Hypothesis: low-dose chest computed tomography, has the same accuracy for the diagnosis of pneumonia compared to the routine protocol. In total, 230 patients are planned to be enrolled in the study.

Each patient will have 2 studies (routine chest CT and low-dose chest CT) sequentially during one visit to the computed tomography room.

DETAILED DESCRIPTION:
As of 30 April 2020, there were over 3 million confirmed cases worldwide, of which over 200,000 were fatal. In Russia at the time of writing, 106 thousand cases of COVID-19 were registered in 78 regions, with 11619 recovered and 1073 dead. Initial prospective analysis of clinical data from 41 patients in Wuhan, with laboratory confirmation of the 2019-nCoV-2 virus, showed that 2019-nCoV-2 caused severe illness, clinically similar to SARS, which sometimes led to the need for hospitalization in the intensive care unit (13 out of 41 [32 %]) and death (6 out of 41 [15%]). All patients with pneumonia in this study had changes in the chest CT scan: preliminary reports indicated that all patients had bilateral lung infiltration.

Given the current prevalence of the disease and the nonspecific symptoms, we expect a significant increase in chest CT scans shortly. A low-dose chest CT scan can be performed with an effective dose of no more than 3.5 mSv, which is much lower than the dose received with a standard protocol - 8-10 mSv.

The investigators hypothesize that a patient with suspected pneumonia can have a low-dose chest CT scan instead of a standard CT while maintaining the accuracy of the method in the diagnosis of inflammatory pulmonary tissue infiltration. The advantage of participating in the study for the patient is the possibility of obtaining an image without motion artifacts that may be associated with coughing, possibly affecting the patient's management tactics.

The study is intended to provide answers to the following questions:

The primary point of the study is to evaluate the correlation between standard CT and low-dose CT scans for the detection of community-acquired pneumonia. The expected correlation percentage is 90%.

The secondary point of study No. 1 is the threshold value of the infiltration zone size detected by low-dose CT scan compared to standard CT scan. Expected threshold - 10 mm.

The secondary point of study No.2 is the number of infiltration zones of pulmonary parenchyma corresponding to viral pneumonia detected by low-dose CT scan in comparison with standard CT scan. Expected number - more than two zones.

In the future, it is planned to use the obtained anonymized data to enter the international registers of images of pneumonia caused by COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* A referral from the attending physician for a chest CT scan
* Suspected pneumonia
* Signed informed consent
* Over 18 years old
* Both male and female

Exclusion Criteria:

* Pregnant or nursing women
* Presence of foreign implanted objects in the body at the scan level (including cardiac pacemakers, spine metalware)
* Patients after surgical intervention at the level of the chest organs
* Cancer patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2020-04-25 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Evaluate the correlation between standard CT and low-dose CT scans for the detection of community-acquired pneumonia. | Upon completion, up to 1 year
  A standardized scale CT1-CT4 will be used. The expected correlation percentage is 90%.

SECONDARY OUTCOMES:
Threshold value of the infiltration zone size detected by low-dose CT scan compared to standard CT scan. | Upon completion, up to 1 year
  Expected threshold - 10 mm.
Number of infiltration zones of pulmonary parenchyma corresponding to viral pneumonia detected by low-dose CT scan in comparison with standard CT scan. | Upon completion, up to 1 year
  Expected number - more than two zones.

CONTACTS AND LOCATIONS:
Locations (1):
- Victor Gombolevskiy, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264